CLINICAL TRIAL: NCT00005546
Title: Molecular Genetic Epidemiology of Three Cardiac Defects -SCOR in Pediatric Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5090; P50HL062178 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Defect, Congenital Heart; Heart Septal Defects, Ventricular; Heart Septal Defects, Atrial; Endocardial Cushion Defects
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Defects, Congenital; Heart Septal Defects, Ventricular; Heart Septal Defects, Atrial; Endocardial Cushion Defects

SUMMARY:
To identify genes involved in the pathogenesis of three types of congenital heart disease, atrial septal defects, paramembranous ventricular septal defects, and atrioventricular canal defects.

DETAILED DESCRIPTION:
BACKGROUND:

Congenital heart defects (CHDs) are thought to result from genetic and environmental factors that disturb cardiac embryogenesis. Because families with multiple members affected with atrial septal defects (ASDs) and atrioventricular canal defects (AVCDs) have been described in previous studies, and the paramembranous ventricular septum is in part completed by the formation of the atrioventricular cushions, this project describes a genetic-epidemiologic study of ASDs, paramembranous ventricular septal defects (VSDs), and AVCDs

DESIGN NARRATIVE:

The study is one of several subprojects within a Specialized Center of Research (SCOR) in Pediatric Cardiovascular Disease. Three groups of subjects, each with surgically- or echocardiographically-confirmed diagnoses of ASDs, VSDs or AVCDs have been identified for study at the University of Iowa Hospitals and Clinics, and at Wolfson Children's Hospital in Jacksonville, Florida. A fourth group of older subjects with ASDs and their progeny will be studied at Iowa because of the reported high recurrence of heart disease in the offspring of subjects with ASDs. The strategy calls upon the molecular genetic capacities available at the University of Iowa to carry out genome-wide searches for genetic loci involved in these defects. Several candidate regions have been identified for ASDs, VSDs and AVCDs. In addition, three well-recognized syndromes provide additional candidate regions - Down syndrome, Holt-Oram syndrome and 8p-syndrome. Parent-affected child trios will be genotyped for closely-spaced markers within these regions and linkage disequilibrium analysis will be used to narrow or exclude these candidate intervals. A genome-wide association study of the trios will employ a parsimonious technique in which DNA from cases with the same CHD phenotype will be pooled, and compared to the pooled DNA from their parents. Loci will be identified where the allele frequency distributions in the affected children and their parents are significantly different. When such loci are identified, a finer localization of the chromosomal area will be undertaken using a high-density set of short tandem repeat polymorphic markers that spans each of the candidate intervals.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Lauer — University of Iowa